CLINICAL TRIAL: NCT03258138
Title: Feasibility and Implementation of a Healthy Lifestyles Program: A Pilot Study
Brief Title: Feasibility and Implementation of a Healthy Lifestyles Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Elizabeth Alvarez, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Healthy lifestyles pilot
Record Dates: First submitted 2017-08-17; First posted 2017-08-23 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Health Behavior; Quality of Life; Chronic Disease; Health Promotion; Stress; Mental Health Wellness 1
Keywords: Pragmatic; Pilot study; Mixed methods; Randomized controlled trial; Implementation research; Person-centered care; Multidisciplinary; Ecological approach
MeSH Terms: conditions — Health Behavior; Chronic Disease | interventions — Health; Exercise

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be allocated to one of the two intervention groups for the duration of the study. One group will be assigned to the more intensive program (MIP= usual care plus healthy lifestyles program) and the other group will be assigned to the less intensive program (LIP= usual care plus health goal development).
Masking Description: The amount of exposure to the programs will be known to participants and providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- More Intensive Program (MIP) (Experimental): Participants will receive the more intensive program, which combines usual care with the full version of the healthy lifestyles program. Participants in this arm will meet weekly for group health and wellness learning sessions or brainstorming group sessions. In addition, they will meet monthly for individual sessions with a multidisciplinary health team, including a family physician, physical therapist and dietician to tailor their health goal development and action plans to their particular needs and situations. They will be asked to maintain physical activity and nutrition journals for a week each every three months.
  Interventions: Behavioral: Health and wellness learning sessions; Behavioral: Brainstorming group sessions; Behavioral: Individual sessions with a multidisciplinary health team; Behavioral: Health goal development; Behavioral: Physical activity and nutrition journals
- Less Intensive Program (LIP) (Experimental): Participants will receive the less intensive program, which combines usual care along with health goal development. Participants in this arm will meet at baseline to set health goals with the support of a research assistant trained in theories of health behaviour and goal setting. They will also meet every three months to measure progress in achieving their goals. They will be asked to maintain physical activity and nutrition journals for a week each every three months.
  Interventions: Behavioral: Health goal development; Behavioral: Physical activity and nutrition journals

INTERVENTIONS:
Behavioral: Health and wellness learning sessions — The health and wellness learning sessions provide a platform for concepts from a variety of health behaviour theories and CBT to be combined with evidence- and practice-based recommendations for healthy lifestyles. They provide the basis for participants' development of an individualized action plan. The sessions will last one hour and participants will receive them in a group setting, 18 times throughout the duration of the program. Specifically, the sessions will be delivered during weeks: 1-8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48.
  Arms: More Intensive Program (MIP)
Behavioral: Brainstorming group sessions — The brainstorming group sessions allow for facilitated discussions where individuals explore barriers and facilitators to achieving their goals and provide an interpersonal component to the program through the building of social interactions. Participants will also receive help in finding community programs to support healthy lifestyles. These sessions will last one hour and participants will receive them in a group setting, 30 times throughout the duration of the program. Specifically, these sessions will be delivered during weeks: 9-11, 13-15, 17-19, 21-23, 25-27, 29-31, 33-35, 37-39, 41-43, 45-47.
  Arms: More Intensive Program (MIP)
Behavioral: Individual sessions with a multidisciplinary health team — Monthly individual sessions with a family physician trained in medical CBT, a dietician and a physical therapist help individuals tailor their action plans and recommendations to their particular circumstances and provide supports based on their needs. The initial session will last 3 hours and occur at baseline. The follow-up sessions will last 1 hour.
  Arms: More Intensive Program (MIP)
Behavioral: Health goal development — Participants in both arms will develop health goals. Several components of these goals will be measured throughout the study, including the stage of change, self-efficacy and actual goal achievement. In the more intensive program arm, participants will develop health goals and learn about how to meet those goals through the group and individual sessions. In the less intensive program arm, participants will receive support in developing health goals from a research assistant trained in theories of health behaviour and in goal setting at baseline, 3 months, 6 months, 9 months and 12 months. The initial goal setting session will be provided within a time period of 2 hours, and the follow-up sessions will be provided within one hour time periods.
Behavioral: Physical activity and nutrition journals — Participants in both arm will be asked to maintain a physical activity journal and a nutrition journal for a week each every three months. These journals help participants reflect on current behaviours and areas for change.

SUMMARY:
Chronic conditions, such as obesity and diabetes, are increasing worldwide. Lifestyle changes (e.g., physical activity, healthy diet, sufficient sleep, managing stress, smoking cessation) are often recommended to prevent or manage these conditions, but changing habits is difficult. Mental health can play a role in the ability to seek out and follow through on the changes necessary to achieve or maintain a healthy lifestyle, yet this aspect is rarely addressed, and access to mental health services is often limited. Furthermore, individuals are influenced by factors at the individual, interpersonal, community and policy levels (e.g., lack of socialization, unsafe neighborhoods). These factors can act as barriers and need to be addressed in order for individuals to make sustainable lifestyle changes.

A new year-long person-centered healthy lifestyles program is proposed to address the "how to" gap in making lifestyle changes through a combination of individual and group sessions. The feasibility and implementation of this new program will be evaluated through a pilot study looking at the full healthy lifestyles program compared to a less intensive version of the program. The study's hypothesis is that the full program will be feasible, acceptable and more effective for helping participants move across stages of change and for meeting their goals than the less intensive program.

DETAILED DESCRIPTION:
A pragmatic mixed methods design including a randomized controlled trial and qualitative components will be used for this pilot study. The randomized controlled trial will include a 1:1 allocation comparing a more intensive program (MIP - usual care plus healthy lifestyles program) with a less intensive program (LIP - usual care plus development of health goals).

The qualitative components include semi-structured interviews of participants (exit interviews at 12 months), MIP staff and participants' healthcare providers (at 6 months and 12 months). In addition, focus groups will be conducted with family members of MIP participants at 9 months. These elements will provide perspectives from multiple stakeholders for improving the healthy lifestyles program and on their roles in creating and maintaining healthy lifestyles.

The primary aim of this study is to assess the feasibility and implementation of the healthy lifestyles program. Impact on participant experiences and outcomes will also be measured. Findings from this study will help inform a larger randomized trial to further look at effectiveness of the program and to determine health system implications. A 2-year extension was approved in order to determine sustainability of findings.

ELIGIBILITY:
Inclusion criteria for randomized controlled trial:

* English-speaking
* 18 years of age or older

Inclusion criteria for qualitative components (family focus groups):

* English-speaking
* 16 years of age or older
* related to participants in randomized controlled trial

Inclusion criteria for qualitative components (program staff):

* Provide services within the more intensive program

Inclusion criteria for qualitative components (healthcare providers):

* Provide health care outside of the healthy lifestyles program for participants in randomized controlled trial

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Retention rates | Baseline to 12 months
  Number of participants recruited and number of participants completing the program

SECONDARY OUTCOMES:
Changes in health goals - Stage of change over time | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  For each health goal, stage of change will be determined with a 7-point Likert scale. Comparisons will be made with baseline but also with other time points.
Changes in health goals - Self-efficacy over time | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  For each health goal, self-efficacy will be determined with a 7-point Likert scale. Comparisons will be made with baseline but also with other time points.
Changes in health goals - Goal achievement over time | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  For each health goal, goal achievement will be determined with a 7-point Likert scale. Comparisons will be made with baseline but also with other time points.
Changes in health-related quality of life on the SF-36 | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  Using a validated scale, health-related quality of life will be measured over time. Comparisons will be made with baseline but also with other time points.
Changes in health-related quality of life on the Health Utilities Index (HUI) 2/3 | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  Using a validated scale, health-related quality of life will be measured over time. Comparisons will be made with baseline but also with other time points.
Changes in the Patient Health Questionnaire (PHQ) | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  Using a validated scale, five common mental health conditions (depression, anxiety, alcohol misuse, somatoform disorder and bulimia) will be measured over time. Comparisons will be made with baseline but also with other time points.
Changes in the Insomnia Severity Index (ISI) | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  Using a validated scale, signs and symptoms of insomnia will be measured over time. Comparisons will be made with baseline but also with other time points.
Changes in the Perceived Stress Scale | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  Using a validated scale, signs and symptoms of perceived stress will be measured over time. Comparisons will be made with baseline but also with other time points.
Changes in the DeJong Gierveld 6-item Loneliness Scale | Baseline, 3 months, 6 months, 9 months and 12 months, 18 months, 24 months, 30 months, 36 months
  Using a validated scale, emotional and social loneliness will be measured over time. Comparisons will be made with baseline but also with other time points.
Changes in blood pressure | Baseline and 12 months, 24 months, 36 months
  Both systolic and diastolic blood pressure will be measured
Changes in weight | Baseline and 12 months, 24 months, 36 months
  Weight will be measured in kilograms
Changes in body mass index (BMI) | Baseline and 12 months, 24 months, 36 months
  Weight and height will be combined to report BMI in kg/m^2
Changes in waist circumference | Baseline and 12 months, 24 months, 36 months
  Measured around waist with a tape measure in inches
Changes in waist:hip ratio | Baseline and 12 months, 24 months, 36 months
  Measured around waist and hips with a tape measure in inches

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Alvarez, MD, MPH, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choban PS, Flancbaum L. The impact of obesity on surgical outcomes: a review. J Am Coll Surg. 1997 Dec;185(6):593-603. doi: 10.1016/s1072-7515(97)00109-9. No abstract available. PMID 9404886
- [Background] Mehrotra C, Remington PL, Naimi TS, Washington W, Miller R. Trends in total knee replacement surgeries and implications for public health, 1990-2000. Public Health Rep. 2005 May-Jun;120(3):278-82. doi: 10.1177/003335490512000310. PMID 16134568
- [Background] El Nakeeb A, Hamed H, Shehta A, Askr W, El Dosoky M, Said R, Abdallah T. Impact of obesity on surgical outcomes post-pancreaticoduodenectomy: a case-control study. Int J Surg. 2014;12(5):488-93. doi: 10.1016/j.ijsu.2014.01.017. Epub 2014 Jan 30. PMID 24486933
- [Background] Liu W, Wahafu T, Cheng M, Cheng T, Zhang Y, Zhang X. The influence of obesity on primary total hip arthroplasty outcomes: A meta-analysis of prospective cohort studies. Orthop Traumatol Surg Res. 2015 May;101(3):289-96. doi: 10.1016/j.otsr.2015.01.011. Epub 2015 Mar 25. PMID 25817907
- [Background] Gibbons CJ, Fournier JC, Stirman SW, DeRubeis RJ, Crits-Christoph P, Beck AT. The clinical effectiveness of cognitive therapy for depression in an outpatient clinic. J Affect Disord. 2010 Sep;125(1-3):169-76. doi: 10.1016/j.jad.2009.12.030. Epub 2010 Jan 18. PMID 20080305
- [Background] Porto PR, Oliveira L, Mari J, Volchan E, Figueira I, Ventura P. Does cognitive behavioral therapy change the brain? A systematic review of neuroimaging in anxiety disorders. J Neuropsychiatry Clin Neurosci. 2009 Spring;21(2):114-25. doi: 10.1176/jnp.2009.21.2.114. PMID 19622682
- [Background] Chesson AL Jr, Anderson WM, Littner M, Davila D, Hartse K, Johnson S, Wise M, Rafecas J. Practice parameters for the nonpharmacologic treatment of chronic insomnia. An American Academy of Sleep Medicine report. Standards of Practice Committee of the American Academy of Sleep Medicine. Sleep. 1999 Dec 15;22(8):1128-33. doi: 10.1093/sleep/22.8.1128. PMID 10617175
- [Background] Resnicow K, DiIorio C, Soet JE, Ernst D, Borrelli B, Hecht J. Motivational interviewing in health promotion: it sounds like something is changing. Health Psychol. 2002 Sep;21(5):444-51. PMID 12211511
- [Background] Sherman MD, Miller LW, Keuler M, Trump L, Mandrich M. Managing Behavioral Health Issues in Primary Care: Six Five-Minute Tools. Fam Pract Manag. 2017 Mar/Apr;24(2):30-35. No abstract available. PMID 28291312
- [Background] Dubord G. Part 1. Goalification. Can Fam Physician. 2010 Dec;56(12):1312. No abstract available. PMID 21375060
- [Background] Dubord G. Part 2. Scalification. Can Fam Physician. 2011 Jan;57(1):54. No abstract available. PMID 21322287
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Patsopoulos NA. A pragmatic view on pragmatic trials. Dialogues Clin Neurosci. 2011;13(2):217-24. doi: 10.31887/DCNS.2011.13.2/npatsopoulos. PMID 21842619
- [Background] Thabane L, Kaczorowski J, Dolovich L, Chambers LW, Mbuagbaw L; CHAP Investigators. Reducing the confusion and controversies around pragmatic trials: using the Cardiovascular Health Awareness Program (CHAP) trial as an illustrative example. Trials. 2015 Sep 2;16:387. doi: 10.1186/s13063-015-0919-3. PMID 26329614
- [Background] Fetters MD, Curry LA, Creswell JW. Achieving integration in mixed methods designs-principles and practices. Health Serv Res. 2013 Dec;48(6 Pt 2):2134-56. doi: 10.1111/1475-6773.12117. Epub 2013 Oct 23. PMID 24279835
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Background] Padwal RS, Pajewski NM, Allison DB, Sharma AM. Using the Edmonton obesity staging system to predict mortality in a population-representative cohort of people with overweight and obesity. CMAJ. 2011 Oct 4;183(14):E1059-66. doi: 10.1503/cmaj.110387. Epub 2011 Aug 15. PMID 21844111
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Marshall D, Pericak D, Grootendorst P, Gooch K, Faris P, Frank C, Bellamy N, Torrance G, Feeny D. Validation of a prediction model to estimate health utilities index Mark 3 utility scores from WOMAC index scores in patients with osteoarthritis of the hip. Value Health. 2008 May-Jun;11(3):470-7. doi: 10.1111/j.1524-4733.2007.00258.x. PMID 18489670
- [Background] Kohrt BA, Luitel NP, Acharya P, Jordans MJ. Detection of depression in low resource settings: validation of the Patient Health Questionnaire (PHQ-9) and cultural concepts of distress in Nepal. BMC Psychiatry. 2016 Mar 8;16:58. doi: 10.1186/s12888-016-0768-y. PMID 26951403
- [Background] Seo JG, Park SP. Validation of the Generalized Anxiety Disorder-7 (GAD-7) and GAD-2 in patients with migraine. J Headache Pain. 2015;16:97. doi: 10.1186/s10194-015-0583-8. Epub 2015 Nov 23. PMID 26596588
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Lynch DJ, McGrady A, Alvarez E, Forman J. Recent life changes and medical utilization in an academic family practice. J Nerv Ment Dis. 2005 Sep;193(9):633-5. doi: 10.1097/01.nmd.0000177778.27069.77. PMID 16131948
- [Background] Reis RS, Hino AA, Anez CR. Perceived stress scale: reliability and validity study in Brazil. J Health Psychol. 2010 Jan;15(1):107-14. doi: 10.1177/1359105309346343. PMID 20064889
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Grygiel P, Humenny G, Rebisz S. Using the De Jong Gierveld Loneliness Scale With Early Adolescents: Factor Structure, Reliability, Stability, and External Validity. Assessment. 2019 Mar;26(2):151-165. doi: 10.1177/1073191116682298. Epub 2016 Dec 8. PMID 27932403
- [Background] Horowitz CR, Robinson M, Seifer S. Community-based participatory research from the margin to the mainstream: are researchers prepared? Circulation. 2009 May 19;119(19):2633-42. doi: 10.1161/CIRCULATIONAHA.107.729863. PMID 19451365
- [Background] Anderson JB. Unraveling health disparities: examining the dimensions of hypertension and diabetes through community engagement. J Health Care Poor Underserved. 2005 Nov;16(4 Suppl A):91-117. doi: 10.1353/hpu.2005.0121. PMID 16327099
- [Derived] Alvarez E, Qutob M, Mbuagbaw L, Lavis J, Lokker C, Walli-Attaei M, Samaan Z, Sutton A, Singh J, Feeny D, Fortuna J. Feasibility and implementation of a healthy lifestyles program in a community setting in Ontario, Canada: protocol for a pragmatic mixed methods pilot study. BMJ Open. 2019 Oct 16;9(10):e031298. doi: 10.1136/bmjopen-2019-031298. PMID 31619429
- See also: Obesity and overweight — http://www.who.int/mediacentre/factsheets/fs311/en/
- See also: Obesity in Canada — http://www.obesitynetwork.ca/obesity-in-canada
- See also: Obesity Puts Young Kids at Risk of Social Isolation — http://www.webmd.com/children/news/20110916/obesity-puts-young-kids-at-risk-of-social-isolation
- See also: Socializing key to "successful aging" — http://www.cbc.ca/news/health/socializing-key-to-successful-aging-1.1260922
- See also: Ontario youth wait a year or more for mental health care: report — https://www.thestar.com/life/health_wellness/2015/05/05/ontario-youth-wait-a-year-or-more-for-mental-health-care-report.html
- See also: Taking patient-centred health care from rhetoric to reality — https://www.theglobeandmail.com/life/health-and-fitness/health/taking-patient-centred-care-from-rhetoric-to-reality/article31077949/
- See also: Maslow's Hierarchy of Needs — https://www.simplypsychology.org/maslow.html
- See also: Prochaska and diclemente's stages of change model - Google Search — https://www.google.ca/search?q=prochaska+and+diclemente%27s+stages+of+change+model&ie=utf-8&oe=utf-8&gws_rd=cr&ei=U__kWM3gDsrqjwTq1ZT4Dg
- See also: Mixed methods embedded design in medical education, mental health and health services research: A methodological analysis — http://digitalcommons.unl.edu/dissertations/AAI3487306
- See also: Chapter 4: Screening for Type 1 and Type 2 Diabetes — http://guidelines.diabetes.ca/browse/chapter4
- See also: HUI Update — https://hqlo.biomedcentral.com/articles/10.1186/1477-7525-1-54
- See also: Measuring and Valuing Health — https://www.sheffield.ac.uk/scharr/sections/heds/mvh/hui2
- See also: Patient Healthcare Questionnaire — http://www.phqscreeners.com/
- See also: Validation of the Insomnia Severity Index as an outcome measure for insomnia research — https://doi.org/10.1016/S1389-9457(00)00065-4

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03258138/Prot_SAP_005.pdf
  • Informed Consent Form: Participants (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03258138/ICF_006.pdf
  • Informed Consent Form: Healthcare providers (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03258138/ICF_007.pdf
  • Informed Consent Form: Program staff (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03258138/ICF_008.pdf
  • Informed Consent Form: Family members (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03258138/ICF_009.pdf